CLINICAL TRIAL: NCT04727047
Title: Neuromuscular Electrical Stimulation for Achilles Tendon Rupture Rehabilitation
Brief Title: NMES for Achilles Tendon Rupture
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment of the number of required patients not completed
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Daniel Cortes, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00016121
Record Dates: First submitted 2020-10-15; First posted 2021-01-27 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Achilles Tendon Rupture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Neuromuscular Electrical Stimulation (Active Comparator): Neuromuscular electrical stimulation will be applied to the calf muscles. The level of stimulation will be increased weekly from 10 to 30 mA during the first 6 weeks after surgery.
  In addition, patients will follow standard therapy for Achilles tendon repair.
  Interventions: Device: neuromuscular electrical stimulation
- Control (No Intervention): Patients will follow standard therapy for Achilles tendon repair.

INTERVENTIONS:
Device: neuromuscular electrical stimulation — All subjects will receive standard rehabilitation for Achilles tendon repair. In addition, neuromuscular electrical stimulation will be applied to the calf muscles of the injured leg. The stimulation volume, the electrode placement and the intensity of the stimulation will be selected based on the mechanical strength of healing Achilles tendon. The intervention will be applied for 6 weeks after repair.
  Arms: Neuromuscular Electrical Stimulation

SUMMARY:
The majority of patients suffering an Achilles tendon rupture develop long term functional deficits in the affected leg. The goal of the proposed study is to evaluate a new rehabilitation protocol using Neuromuscular Electrical Stimulation (NMES) for reducing muscle atrophy and improving tendon properties. If proven beneficial, the proposed protocol can be easily adopted and incorporated as part of routine care for Achilles tendon rupture.

DETAILED DESCRIPTION:
Achilles Tendon Ruptures (ATR) are common and permanently affect the function of the lower leg. Regardless of treatment approach the majority of patients develop long term functional deficits, which include decreased plantar flexion strength, lower heel-rise height, and altered gait patterns. It is believed that tendon lengthening and calf muscle atrophy, which develop during the first few weeks of recovery, are major factors contributing to these functional deficits. The initial development of atrophy is likely caused by reduced loading and muscle activity of the affected leg. However, long-term atrophy may be related to tendon elongation. On the other hand, tendon elongation initially rises during the first few weeks of unloading and slowly reduces, but not completely, when loading is resumed. However, atrophied calf muscles may not provide sufficient loading for optimal tendon recovery. Therefore, there seems to be vicious spiral between tendon elongation and muscle atrophy.

The objective of this study is to develop a neuromuscular electrical stimulation (NMES) rehabilitation protocol for Achilles tendon ruptures. Our preliminary data has shown that force applied to the tendon can be modulated using electrical intensity and pad placement. Therefore, NMES can produce significant contraction in the calf muscles and induce controllable, low-magnitude, cyclic loading to the tendon; which cannot be achieved with voluntary muscle contractions. This approach can potentially overcome limitations of the current rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Achilles tendon rupture

Exclusion Criteria:

1. Those unable to understand spoken English.
2. Participants treated non-operatively
3. Augmented surgical repair (i.e., use of additional tissue at the repair site)
4. Tendon ruptures associated with the use of fluoroquinolones (Examples include ciprofloxacin (Cipro), gemifloxacin (Factive), levofloxacin (Levaquin), moxifloxacin (Avelox), norfloxacin (Noroxin), and ofloxacin (Floxin))
5. Allergy to ultrasound gel
6. Any other condition affecting the ability of the participant to walk or jump
7. Any other health conditions known to impair normal healing: Diabetes, Cardiovascular conditions decreasing blood supply to the leg
8. Those unable to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Ability to perform a single heel rise | Week 12
  The ability of patients to perform a single heel rise using the injured will be tested.

SECONDARY OUTCOMES:
Tendon length | Week 6 and12
  Length from the tendon insertion to the myotendinous junction
Tendon cross-sectional area | Week 6, 12
  Area of the tendon measured via ultrasound imaging at the rupture location
Gastrocnemius muscle cross-sectional area | Week 1, 6, 12
  Area of the tendon measured via ultrasound imaging at the rupture location
Soleus muscle cross-sectional area | Week 1, 6, 12
  Area of the tendon measured via ultrasound imaging at the rupture location
Foot and Ankle Outcome Score (FAOS) | Week 6, 12
  Score that assesses patient pain, other symptoms, function in daily living, function in sport and recreation, and foot/ankle related quality of life. Scores range from 0 to 100 with a score of 0 indicating the worst possible foot/ankle symptoms and 100 indicating no foot/ankle symptoms.
Achilles Total Rupture Score | Week 6, 12
  It consists of ten items evaluating aspects of symptoms and function. Each item has scores ranging between 0 and 10 on a Likert scale. The instrument therefore has a maximum score of 100, which corresponds to no symptoms and full function.
Tampa Scale for Kinesiophobia (TSK) | Week 6, 12
  Questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. The total score of the scale range from 17- 68, where 17 means no kinesiophobia, 68 means severe kinesiophobia, and score ± 37 indicates there is kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State University, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT04727047/Prot_SAP_000.pdf